CLINICAL TRIAL: NCT03091517
Title: A Single Arm Feasibility Study of GlycoLeap, an On-line Lifestyle Modification and Self-management Program for People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GlycoLeap
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Online lifestyle modification; Self-management; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GlycoLeap (Other): Since this is a single arm study, all participants will receive the GlycoLeap intervention.
  Interventions: Behavioral: GlycoLeap

INTERVENTIONS:
Behavioral: GlycoLeap — GlycoLeap is a 24-week programme includes the following features:
  Interactive Education Lessons: Beginning week 1, the participant will be presented with a diabetes self-management education curriculum. These lessons are divided into 6 phases, and each lesson is fully accessible online from a computer or mobile phone, and takes approximately 10 - 15 minutes to complete.
  The Glyco Mobile Application: During the 24 week intervention period, the participant will use the Glyco mobile application that allows them to track their weight (measured on the wireless weighing scale), self-tested glucose readings (measured using the glucometer kit), and log their foods and meals by taking photos using their phone. A health coach will review the participant's data regularly, provide personalised feedback.

SUMMARY:
This single arm pilot study will explore the feasibility of GlycoLeap, a proprietary online lifestyle modification and self-management education program developed in Singapore for people with type 2 diabetes, as an add-on to primary care delivered through one of the SingHealth Polyclinics.

DETAILED DESCRIPTION:
Lifestyle modification - focusing on a healthy diet, regular exercise and behaviour change - are the mainstay of first-line therapies in managing diabetes. There is strong evidence that lifestyle interventions can result in modest weight loss and improvements in clinical metrics such as glycated haemoglobin (HbA1c), blood pressure and cholesterol. For people with type 2 diabetes, lifestyle modification and self-management education can lead to improved clinical outcomes and reduced risks of complications.

Operationally, such interventions are often difficult to administer in the primary care and community setting because of lack of provider time/resources/training and difficulty in engaging patients. Fortunately, there is a growing body of evidence which shows that online programs and smartphone-based interventions can lead to improved clinical outcomes like weight loss and HbA1c reduction. Moreover, these interventions can be disseminated to a larger group of people and at a low cost. However, results from community based studies often fail to live up to what is achieved in clinical trials due to lack of clinician oversight and support. Without this support, patients often fail to engage in the intervention to the levels required for health benefits to materialize.

This feasibility study will explore the use of GlycoLeap, a proprietary online lifestyle modification and self-management education program developed in Singapore for people with type 2 diabetes, as an add-on to primary care delivered through one of the SingHealth Polyclinics. The goal of the study is to test whether patients with diabetes who receive care at the clinic are amenable to such an intervention, to quantify program fidelity for those who do enroll in the study, and to explore the extent to which the intervention can be used in conjunction with primary care in efforts to improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 - 70 years
2. Medical diagnosis of Type 2 diabetes in electronic health records or based on World Health Organisation diagnostic criteria
3. Last HbA1c result within 2 months of ≥ 7.5%
4. BMI > 23 kg/m2 (if Asian) or BMI > 25 kg/m2 (if non-Asian)
5. Not on insulin
6. Owns a smartphone (iPhone or Android phone) and able to use it

Exclusion Criteria:

1. Last HbA1c blood test older than 2 months
2. Cancer requiring treatment in past 5 years
3. Cardiovascular disease (heart attack or cardiac procedure within past 3 months)
4. Stroke or history/treatment for transient ischemic attacks in past 3 months
5. Chronic renal failure or dialysis
6. Amputation of lower limbs
7. Current use of medication for weight loss
8. Chronic treatment with systemic corticosteroids
9. History of bariatric surgery or extensive bowel resection
10. Unable to understand English

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels (Effectiveness) | Baseline, Month 6
  HbA1c or glycated haemoglobin is a measure of blood glucose levels. We will assess change in HbA1c levels.

SECONDARY OUTCOMES:
Change in weight (Effectiveness) | Baseline, Month 6
  We will assess change in weight
Proportion of individuals who are willing to participate (Reach) | Baseline
  Percentage of participants offered the GlycoLeap programme who agree to enrol
Extent of engagement in completing online health lessons (Implementation) | Throughout 6 month intervention duration
  Number of online GlycoLeap health lessons completed
Extent of engagement in submitting blood glucose logs (Implementation) | Throughout 6 month intervention duration
  Number of blood glucose measurements logged per week in GlycoLeap's smartphone app
Extent of engagement in submitting weight logs (Implementation) | Throughout 6 month intervention duration
  Number of weight measurements logged per week in GlycoLeap's smartphone app
Extent of engagement in submitting meal logs (Implementation) | Throughout 6 month intervention duration
  Number of meals logged per week in GlycoLeap's smartphone app
Extent of engagement with health coach (Implementation) | Throughout 6 month intervention duration
  Number of messages sent to health coaches per week through GlycoLeap's smartphone app
Change in HbA1c (primary outcome) as a function of program engagement (Effectiveness) | Baseline, Month 6, Throughout 6 month intervention duration
  We will test whether those with greater engagement with the GlycoLeap program show greater improvements in HbA1c (primary outcome).
Change in weight loss (secondary outcome) as a function of program engagement (Effectiveness) | Baseline, Month 6, Throughout 6 month intervention duration
  We will test whether those with greater engagement with the GlycoLeap program show greater improvements in weight loss (secondary outcome).
Degree of user satisfaction with the GlycoLeap program (Maintenance) | Month 6
  We will conduct a preliminary assessment of maintenance at the individual level via a user satisfaction survey at the month 6 follow-up. Participants will rate the smartphone app on a scale of 1 (Poor) to 5 (Excellent) and whether they would recommend the app to others for managing their diabetes on a scale of 1 (Would not recommend) to 5 (Would highly recommend).

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Polyclinics - Tampines, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Koot D, Goh PSC, Lim RSM, Tian Y, Yau TY, Tan NC, Finkelstein EA. A Mobile Lifestyle Management Program (GlycoLeap) for People With Type 2 Diabetes: Single-Arm Feasibility Study. JMIR Mhealth Uhealth. 2019 May 24;7(5):e12965. doi: 10.2196/12965. PMID 31127720